CLINICAL TRIAL: NCT06800313
Title: Phase 1/2 Study of HLD-0915 in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: A Study of HLD-0915 in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Halda Therapeutics OpCo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HLD-0915-ONC-101
Record Dates: First submitted 2025-01-20; First posted 2025-01-30 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer Metastatic Disease; Prostate Cancer (Adenocarcinoma)
Keywords: prostate cancer; RIPTAC; HLD-0915
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Phase 1 dose escalation will employ the BF-BOIN design (to find the Maximum Tolerated Dose (MTD)/ Recommended Dose for Expansion (RDE). BF-BOIN enables backfilling patients to doses that are cleared for safety during the dose escalation, thereby generating additional data on safety, tolerability, and preliminary activity on doses below the MTD. This facilitates the identification of the RDE(s). The BF-BOIN consists of two interrelated components: dose escalation and backfill.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HLD-0915 (Experimental): Oral HLD-0915 administered as a single agent on a 21-day treatment cycle.
  Interventions: Drug: HLD-0915

INTERVENTIONS:
Drug: HLD-0915 — A treatment cycle consists of 21 days. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.)

SUMMARY:
Assessment of the safety and efficacy of HLD-0915 as monotherapy in patients with metastatic castration resistant prostate cancer (mCRPC) that have progressed on prior systemic therapies, once a recommended dose for expansion (RDE) has been determined in Phase 1 of the trial.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label study of the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and anti-tumor activity of oral single-agent HLD-0915. Patients on the study must continue androgen deprivation therapy (ADT) unless surgically castrated,

The study will include an initial Phase 1 portion to determine the maximum tolerated dose (MTD) and/or recommended dose(s) for expansion (RDEs) of HLD-0915 as monotherapy and Phase 2 expansion cohorts to further evaluate the efficacy and safety of HLD-0915.

Phase 1 of this study is an open-label, dose-escalation and cohort expansion study in patients with mCRPC that have progressed after prior systemic therapies. Patients will be enrolled in monotherapy dose-escalation cohorts using a Bayesian optimal interval with backfill (BF-BOIN) design. Patients are treated in cohort size of 3 with the enrollment staggered between cohorts.

Phase 2 of this study will evaluate the anti-tumor activity of HLD-0915 administered at the RDEs in patients with mCRPC. Phase 2 study design and patient population will be based on the outcomes of Phase 1 of the trial.

ELIGIBILITY:
Key Inclusion Criteria:

All patients must meet the following criteria to be eligible for Phase 1 study participation:

1. Males of age 18 years at the time of signing the informed consent form (ICF).
2. Able to understand and voluntarily sign an informed consent document prior to any study-related assessments/procedures.
3. Patients must have histological, pathological, and/or cytological confirmation of adenocarcinoma of the prostate.
4. Patients must have prior orchiectomy and/or ongoing androgen-deprivation therapy and a castrate level of serum testosterone.
5. Patients must have progressed on prior line(s) of therapy.
6. Patients must have progressive mCRPC defined as having demonstrated PSA progression on the prior regimen. PSA progression may have occurred with or without accompanying radiographic progression.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
8. Life expectancy of at least 3 months.
9. Adequate hematological, renal, and hepatic function.
10. Able to swallow an oral medication.
11. Willing and able to adhere to the study visit schedule and other protocol requirements.
12. Patients on a stable bisphosphonate or denosumab regimen for 30 days prior to enrollment are eligible.

Key Exclusion Criteria:

Patients with any of the following will be excluded from participation in Phase 1 of the study:

1. Has experienced a recent major bleed or has a known bleeding disorder.
2. Tumors exhibiting neuroendocrine or small cell carcinoma component by histopathology.
3. Receiving continuous corticosteroids at prednisone-equivalent dose of >10 mg/day.
4. Has received systemic anti-cancer therapy (cytotoxic chemotherapy, biologic agent, checkpoint inhibitors, or radiation therapy) or investigational drugs within 2 weeks prior to first dose of study drug with certain exceptions requiring longer washout periods.
5. History of myocardial infarction or unstable angina within 6 months prior to enrollment, or clinically significant cardiac disease.
6. Known clinically significant active or chronic infection.
7. Acute or chronic uncontrolled renal disease, pancreatitis, or liver disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Frequency of dose-limiting toxicities (DLTs) | 21 days
Phase 1: Frequency and severity of AEs and serious adverse events (SAEs), including abnormal clinical observations, abnormal ECG parameters, abnormal laboratory assessments and abnormal vital signs changed from baseline | 21 days

SECONDARY OUTCOMES:
Phase 1: Plasma concentrations of HLD-0915 as a function of time post-dosing | 21 days
Phase 1: Plasma PK Parameters (Cmax) | 21 days
  Maximal plasma concentration of HLD-0915
Phase 1: Plasma PK Parameters (Tmax) | 21 days
  Time to maximal plasma concentration of HLD-0915
Phase 1: Plasma PK Parameters (T1/2) | 21 days
  Plasma half-life of HLD-0915
Phase 1: Plasma PK Parameters (AUC0-inf) | 21 days
  Plasma area under the curve of HLD-0915
Phase 1: The proportion of pts with a confirmed prostate-specific antigen (PSA) decline ≥30%, ≥50%, and ≥90% | 21 days
Phase 1: Objective response rate (ORR) per RECIST in evaluable patients | 21 days
Phase 1: Duration of response (DOR) | 21 days
Phase 1: Radiographic progression-free survival (rPFS) | 21 days
Phase 1: Time to response (TTR) | 21 days
Phase 1: Change in PSA over time | 21 days

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Yale - New Haven Hospital - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists, Sarasota, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - START Midwest, LLC, Grand Rapids, Michigan
  - Evelyn H. Lauder Breast and Imaging Center (BAIC), New York, New York
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - SCRI Oncology Partners, Nashville, Tennessee
  - NEXT Austin, Austin, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No